CLINICAL TRIAL: NCT03427606
Title: Laparoscopic Sacral Colpopexy for Pelvic Organ Prolapse: Continuous Suture for Mesh Fixation
Brief Title: Continuous Locked Non-barbed Suture for Mesh Fixation During Laparoscopic Sacral Colpopexy for Severe Pelvic Organ Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Principal Investigator, Andrea Morciano, M.D., Azienda Ospedaliera Cardinale G. Panico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSCContinua
Record Dates: First submitted 2018-01-30; First posted 2018-02-09 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: sacral colpopexy; laparoscopy; mesh fixation
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Suture (Experimental)
  Interventions: Procedure: Continuous Locked Suture vs Traditional 5-points suture for Laparoscopic Sacral Colpopexy
- Single 5-points Suture (Active Comparator)
  Interventions: Procedure: Continuous Locked Suture vs Traditional 5-points suture for Laparoscopic Sacral Colpopexy

INTERVENTIONS:
Procedure: Continuous Locked Suture vs Traditional 5-points suture for Laparoscopic Sacral Colpopexy — To verify if the operative time of a standard laparoscopic sacral colpopexy associated to subtotal hysterectomy for the treatment of POP could be further reduced using continuous locked suture vs traditional 5-points suture for mesh fixation

SUMMARY:
This prospective randomized pilot study is aimed to verify if the operative time of a standard laparoscopic sacral colpopexy associated to subtotal hysterectomy for the treatment of POP could be further reduced using a continuous locked suture vs. conventional single 5-points suture for anterior mesh fixation.

DETAILED DESCRIPTION:
Introduction Pelvic-organ prolapse, in which the pelvic organs (uterus, bladder, and bowel) protrude into or past the vaginal introitus, is a condition often treated with surgery. Women have an 11 percent risk of surgery for prolapse or urinary incontinence by 80 years of age, and of this 11 percent, almost one third of the women have a second surgery. This fact points to the need for improved treatment of pelvic-floor disorders. Numerous surgical procedures have been described for the management of POP. Vaginal surgery may be associated with less postoperative pain and a more rapid return to daily living than abdominal repair. However, in a randomised study, sacrocolpopexy was twice as likely to result in optimal anatomical outcome as vaginal surgery. Laparoscopic sacrocolpopexy provides the potential to combine the success rates of an abdominal approach with the faster recovery associated with a minimally invasive technique. Tissue dissection and mesh placement may also be facilitated by the magnification and field of view permitted by the laparoscopic approach. These benefits must be balanced against a longer operating time from 150 to 250 minutes according to surgeons' experience. In addition, this procedure is often associated to subtotal hysterectomy (LSH) for the reasons of prevention (post-menopause age) or uterine diseases, which improve still more the operating time.

This prospective randomized pilot study is aimed to verify if the operative time of a standard laparoscopic sacral colpopexy associated to subtotal hysterectomy for the treatment of POP could be further reduced using using a continuous locked suture vs. conventional 5-points single suture for anterior mesh fixation.

Secondary endopoints of this comparison are incidence of intra- or postoperative complications estimated blood loss, postoperative pain (evaluated by VAS), days of hospitalization and costs for the health care system.

Statistical Analysis and Study Design This is a single Institution prospective randomized clinical trial conducted at the Pia Fondazione Panico of Tricase, Italy.

To have an imbalanced results and to reduce any bias, a randomization list has been checked.

Probability (p) values will be considered to be statistically significant at the <0.05 level.

There will be recruited 20 patients to treat using continuous locked suture and 20 patients to treat with standard 5-points single suture for mesh fixation comparing these two techniques in terms of operative time, estimated blood loss and other intra- or post operative complications, postoperative pain, days of hospitalization, costs. All patients will be adequately informed and inserted in the study only after having read and signed an informed consent. Diagnostic, clinical and surgical data of each patient will be prospectively recorded. At the end of the procedure, a schedule will be compiled with intraoperative data. All clinical and histologic data will be recorded prospectively using a database. Pain associated with the procedure will be evaluated by a subjective assessment (analysis of VAS scale values reported by patients at 8 and 24 hours after surgery). Post-operative complications will be evaluated during the first 30 days after surgery according to Dindo's classification.

ELIGIBILITY:
Inclusion Criteria:

For patients

* Age ≤ 80 years
* Patient's informed consent
* American Society of Anesthesiologists: < class III or IV
* Physiologic, surgical or iatrogenic menopause.
* No previous major abdominal surgical procedures

For diseases

* POP-Q stage III/IV for anterior and/or apical compartment; stage <III for posterior compartment.
* No uterine cervix dysplasia or endometrial disorders.
* No uterine size larger than conform 10 weeks gestation

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Operative Time | through study completion, an average of 1 year
  Operative time for LPS subtotal hysterectomy and sacral colpopexy operative time will be calculated from the entrance in the abdominal cavity.

SECONDARY OUTCOMES:
Recurrent Prolapse | through study completion, an average of 1 year
  Appearance of recurrent prolapse after one year from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morciano, M.D., Principal Investigator — Pia Fondazione Giovanni Panico